CLINICAL TRIAL: NCT03520101
Title: Comparison of the Balloon-Expandable Edwards Valve and Self-Expandable CoreValve Evolut R or Evolut PRO System for the Treatment of Small, Severely Dysfunctional Surgical Aortic Bioprotheses: A Pilot Prospective Randomized Trial. The 'LYTEN' Trial
Brief Title: Comparison of the Balloon-Expandable Edwards Valve and Self-Expandable CoreValve Evolut R or Evolut PRO System for the Treatment of Small, Severely Dysfunctional Surgical Aortic Bioprotheses. The 'LYTEN' Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, Principal investigator, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LYTEN
Record Dates: First submitted 2017-05-08; First posted 2018-05-09 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Aortic Valve Stenosis; Regurgitation, Aortic; Prosthesis Failure
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency; Prosthesis Failure

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized trial including patients with surgical aortic bioprosthetic dysfunction in the presence of a small stented surgical valve. Patients will be randomized to either receive an Edwards (SAPIEN XT or SAPIEN 3) valve or a Core Valve Evolut R or Evolut PRO system.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAPIEN (Other): Following the Heart Team's decision to proceed with a TAVI-ViV procedure, patients will received an Edwards (SAPIEN XT or SAPIEN 3) valve.
  Interventions: Procedure: TAVI_ViV procedure with Edwards valve
- COREVALVE (Other): Following the Heart Team's decision to proceed with a TAVI-ViV procedure, patients will received the CoreValve Evolut R or Evolut PRO valve system.
  Interventions: Procedure: TAVI_ViV procedure with CoreValve system

INTERVENTIONS:
Procedure: TAVI_ViV procedure with Edwards valve — The TAVR procedure will be performed following the standards of each participating center. No restriction or specific recommendation will be given regarding the approach, general vs. local anesthesia, imaging guidance during the TAVI procedure, and post-procedural TAVI management. The decision for selecting either a 20 or 23mm Edwards valve will be based on 3D CT measurements of the mean inner diameter of the surgical aortic bioprosthesis. A 23mm Sapien 3 valve will be recommended if the inner diameter is >18 mm, and a 20mm valve will be selected if the mean inner diameter is ≤18 mm.
  Arms: SAPIEN
Procedure: TAVI_ViV procedure with CoreValve system — The TAVR procedure will be performed following the standards of each participating center. No restriction or specific recommendation will be given regarding the approach, general vs. local anesthesia, imaging guidance during the TAVI procedure, and post-procedural TAVI management. A 23mm valve will be recommended in all patients randomized to the self-expanding CoreValve Evolut R system.
  Arms: COREVALVE

SUMMARY:
The treatment with transcatheter aortic valve implantation (TAVI) of patients with small (≤23mm) surgical bioprostheses remains a challenge due to the increased transvalvular residual gradients and high rates of severe prosthesis-patient mismatch (PPM) following the procedure.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized open-label trial including patients with surgical aortic bioprosthetic dysfunction in the presence of a small (≤23mm; inner diameter ≤21 mm) stented surgical valve. Following the Heart Team'S decision to proceed with a TAVI-ViV procedure, patients will be randomized to either receive an Edwards (SAPIEN XT or SAPIEN 3) valve or a CoreValve Evolut R or Evolut PRO system. New iterations of these valve models may also be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients with surgical aortic bioprosthetic dysfunction defined as severe aortic stenosis and/or regurgitation approved for a ViV procedure by the Heart Team
* Stented surgical valves.
* Small (≤23mm) surgical valve

Exclusion Criteria:

- Stentless or sutureless surgical valves

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of prothesis-patient mismatch (PPM) (valve performance) | 30 days
  Severe prothesis-patient mismatch (PPM) (defined as an index aortic valve area ≤0.65 cm2/m2) and/or moderate-severe aortic regurgitation (AR) (VARC-2 definition).
Residual transvalvular gradient | 30 days
  Residual (maximal and mean) transvalvular gradient.

SECONDARY OUTCOMES:
Transvalvular gradient. | 1-year
  Maximal and mean transvalvular gradient
Valve performance : Moderate or severe PPM moderate-severe AR at 30 days and 1 year. | 30 days and 1 year
  Moderate or severe PPM; moderate-severe AR.
Combined endpoints: Moderate-severe AR or severe PPM at 1-year follow-up. | 1 year
  Moderate-severe AR or severe PPM.
Clinical safety endpoints | 30 days and 1 year
  individually and combined: death, stroke, major or life threatening bleeding, pacemaker implantation, myocardial infarction.
Exercise capacity | 30 days and 1 year
  Exercise capacity as evaluated by the six-minute walk test
Changes in LV hypertrophy | 30 days and 1 year
  Changes in LV hypertrophy

CONTACTS AND LOCATIONS:
Overall Officials: Josep Rodés-Cabau, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- IUCPQ, Québec, Canada

REFERENCES:
- [Derived] Cepas-Guillen P, Abbas AE, Serra V, Vilalta V, Nombela-Franco L, Regueiro A, Al-Azizi KM, Iskander A, Conradi L, Forcillo J, Lilly S, Calabuig A, Fernandez-Nofrerias E, Mohammadi S, Giuliani C, Pelletier-Beaumont E, Pibarot P, Rodes-Cabau J. Balloon- Versus Self-Expanding Transcatheter Valves for Failed Small Surgical Aortic Bioprostheses: 3-Year Results of the LYTEN Trial. Circ Cardiovasc Interv. 2026 Feb 2:e016255. doi: 10.1161/CIRCINTERVENTIONS.125.016255. Online ahead of print. PMID 41623058
- [Derived] Nuche J, Abbas AE, Serra V, Vilalta V, Nombela-Franco L, Regueiro A, Al-Azizi KM, Iskander A, Conradi L, Forcillo J, Lilly S, Calabuig A, Fernandez-Nofrerias E, Mohammadi S, Giuliani C, Pelletier-Beaumont E, Pibarot P, Rodes-Cabau J. Balloon- vs Self-Expanding Transcatheter Valves for Failed Small Surgical Aortic Bioprostheses: 1-Year Results of the LYTEN Trial. JACC Cardiovasc Interv. 2023 Dec 25;16(24):2999-3012. doi: 10.1016/j.jcin.2023.10.028. Epub 2023 Oct 23. PMID 37902146
- [Derived] Rodes-Cabau J, Abbas AE, Serra V, Vilalta V, Nombela-Franco L, Regueiro A, Al-Azizi KM, Iskander A, Conradi L, Forcillo J, Lilly S, Calabuig A, Fernandez-Nofrerias E, Mohammadi S, Panagides V, Pelletier-Beaumont E, Pibarot P. Balloon- vs Self-Expanding Valve Systems for Failed Small Surgical Aortic Valve Bioprostheses. J Am Coll Cardiol. 2022 Aug 16;80(7):681-693. doi: 10.1016/j.jacc.2022.05.005. Epub 2022 May 18. PMID 35597385